CLINICAL TRIAL: NCT05264545
Title: Prospective, Multicenter, Non-randomized, Controlled Clinical Study Utilizing Non-Guided vs. Guided Surgery to Immediately Loaded PrimeTaper Implants in Partially Edentulous Patients
Brief Title: Non-Guided vs. Guided Surgery to Immediately Loaded PrimeTaper Implants in Partially Edentulous Patients
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: McGuire Institute (Industry)
Collaborators: Dentsply Sirona Implants and Consumables (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DS2021-01
Record Dates: First submitted 2021-09-24; First posted 2022-03-03 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Partially Edentulous Maxilla or Mandible

STUDY DESIGN:
Intervention Model Description: Prospective, multicenter, non-randomized, controlled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Single Arm (Other): There are no arms in the study, it is a non randomized, controlled study
  Interventions: Device: PrimeTaper EV

INTERVENTIONS:
Device: PrimeTaper EV — The PrimeTaper EV Implant is a screw shaped dental implant with a defined surface achieved through grit blasting, followed by a process involving a treatment in diluted hydrofluoric acid. There is a conical connection between the implants and the abutments for a tight and stable connection.

SUMMARY:
A 510k approved dental device for subjects requiring single or multiple tooth replacement with implants where immediate restoration/loading is preferred.

DETAILED DESCRIPTION:
The rationale for this study is to provide scientific data on the clinical performance and patient reported outcomes of the PrimeTaper EV implant when utilizing non-guided vs guided surgical technique. The PrimeTaper EV implant has the OsseoSpeed surface, which is especially indicated for use in soft bone applications where implants with other surface treatments may be less effective.

The main interests of this study are to assess the survival and the success rates of the implants supporting maxillary or mandibular fixed single or 2-fixture restorations after 1, 2, 3, 4 and 5 years in function

ELIGIBILITY:
Inclusion Criteria:

1. Subject ≥25 years.
2. Subject has signed and dated the informed consent form prior to any study procedures.
3. History of either a healed edentulous area or single or multiple teeth requiring extraction and in need of a single or fixed bridge prosthetic restoration and where immediate restoration/loading is preferred.
4. Opposing jaw in the treatment area meets any of the following stable occlusal conditions:

Complete denture Partial removable denture Fixed bridges and/or crowns Natural dentition

Exclusion Criteria:

Any of the following is regarded as a criterion for exclusion from the study (all criteria apply at study inclusion, but criteria numbered 1-4 also apply during the entire study period):

1. Unlikely to be able to comply with study procedures, according to the Investigator's judgment.
2. Subject is not willing to participate in the study or not able to understand the content of the study.
3. Involved in the planning and conduct of the study.
4. Unable or unwilling to return for follow-up visits for a period of 5 years.
5. Has an uncontrolled pathological process in the oral cavity (e.g. untreated periodontal disease, uncontrolled caries, severe malocclusion, etc.).
6. Known or suspected current malignancy.
7. History of radiation therapy in the head and neck region.
8. History of chemotherapy within 5 years prior to surgery.
9. Systemic or local disease or condition that could compromise post-operative healing and/or osseointegration (e.g., uncontrolled diabetes mellitus as reported by the subject).
10. Use of systemic corticosteroids, IV bisphosphonates or any other medication that could compromise post-operative healing and/or osseointegration.
11. Current alcohol and/or drug abuse.
12. Smoking more than 10 cigarettes of any type per day.
13. Current need for major bone grafting and/or augmentation in the planned implant area (esthetic augmentation and minor facial grafting are allowed).
14. Known pregnancy, or plans to become pregnant during the study period of 5 years
15. Participation in another clinical study within the previous 6 months that may interfere with the present study.

    Post-surgical Exclusion criteria
16. Insufficient primary stability, as judged by the investigator, of the implant(s).
17. Severe non-compliance to CIP as judged by the Investigator and/or Dentsply Sirona Implants.

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2022-03-22 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
To evaluate implant survival rate at 1 year after final restoration attachment (screw retained when feasible) with single and multiple (fixed bridges) PrimeTaper EV implant(s) utilizing non-guided versus guided surgery | 1 year after final restoration
  Number of remaining implants counted clinically and radiographically, i.e. 'Yes' or 'No' for each implant where 'Yes' means that the implant is still remaining and 'No' means that the implant is not remaining.

SECONDARY OUTCOMES:
Implant stability by manual clinical examination | throughout study, up to the 5 year follow up
  Mobility (manual stability) will be assessed by a percussion test for resonance indicative of bone to implant contact vertically and laterally.
Implant survival rate | 2, 3, 4, and 5 years after final restoration attachment
  Number of remaining implants counted clinically and radiographically, i.e. 'Yes' or 'No' for each implant where 'Yes' means that the implant is still remaining and 'No' means that the implant is not remaining.
Maintenance of marginal bone levels on patient- and implant level. | throughout study up to the 5 year follow up visit
  Changes (mm) in marginal bone level (MBL)
Condition of the peri-implant mucosa (Plaque Index) | measured at 12 days (no BOP, PPD), 16 weeks, 20 weeks, 6 months, 1,2,3,4,5 years,
  Plaque index will be measured following implant placement by visual inspection using a scoring system of 0-1, 0 being no plaque is present and 1 being plaque is present.
Condition of the peri-implant mucosa (Recession) | measured at 12 days (no BOP, PPD), 16 weeks, 20 weeks, 6 months, 1,2,3,4,5 years,
  Recession will be measured following implant placement by placing a probe between the tooth and gum to record depth of recession in millimeters from the crown margin to the gingival margin rounded to the nearest 0.5 mm.
Condition of the peri-implant mucosa (Suppuration by visual inspection). | measured at 12 days (no BOP, PPD), 16 weeks, 20 weeks, 6 months, 1,2,3,4,5 years,
  Suppuration presence or absence will be measured following implant placement by using a scoring system of 0-1. 0 being no suppuration and 1 being suppuration is present. It is being identified by visual inspection and palpitation of moderate inflammation.
Condition of the peri-implant mucosa. | measured at 12 days, 20 weeks, 1,2,3,4,5 years
  Keratinized Tissue Width (KTw) will be measures following implant placement
Patient Reported Outcomes (PROs) | 20 weeks, 6 months, years 1,2,3,4,5
  subjects will be interviewed to ask about Discomfort using a 0 (no discomfort)-10 (as much discomfort as i have ever felt) point grading system
Patient Reported Outcomes (PROs) | 20 weeks, 6 months, years 1,2,3,4,5
  subjects will be interviewed to ask about Esthetics using a 0 (completely displeased)-10 (completely pleased) point grading system
Patient Reported Outcomes (PROs) | 20 weeks, 6 months, years 1,2,3,4,5
  subjects will be interviewed to ask about Satisfaction using a 0 (completely dissatisfied) -10 (completely satisfied) point grading system
Investigator Assessment of the Implant-Prosthetic Complex | 20 weeks and 5 years.
  Evaluation of the Esthetic outcome on a 4 point scale (1=very good, 2= good, 3=acceptable, 4=not acceptable)
Investigator Assessment of the Implant-Prosthetic Complex | 20 weeks and 5 years.
  Evaluation of Function a 4 point scale (1=very good, 2= good, 3=acceptable, 4=not acceptable)
Investigator Assessment of the Implant-Prosthetic Complex | 20 weeks and 5 years.
  Evaluation of Gingival Health n a 4 point scale (1=very good, 2= good, 3=acceptable, 4=not acceptable)
Investigator Assessment of the Implant-Prosthetic Complex | 20 weeks and 5 years.
  Evaluation of Bone Level of the permanent prosthetic restoration n a 4 point scale (1=very good, 2= good, 3=acceptable, 4=not acceptable)
Implant success | throughout study up to the 5 year follow up visit
  Proportion of implants with the derived answer 'No' on the occurrence of "pain", "mobility", "≥2 mm radiological bone loss from initial placement", "infection", "radiolucency" and "6" or greater on the Subject Satisfaction PRO Question and "Very good", "good" or "acceptable" on each Investigator Evaluation of Esthetic Outcome, Function, Gingival Health, Bone Level
Prosthetic survival | 5 years after final restoration attachment
  Proportion of original permanent prosthetic restorations still in place at the 5 years after final restoration attachment.
Prosthetic success | 5 years after final restoration attachment.
  Analysis of successful permanent prosthetic restorations (implant-prosthetic complex); Number of suprastructure fractures, technical repairs 5 years after final restoration attachment.

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - McClain and Schallhorn Periodontics and Implant Dentistry, Aurora, Colorado
  - Colorado Gum Care, Broomfield, Colorado
  - Periodontal Medicine Surgical Specialists, LLC, Oakbrook Terrace, Illinois
  - Metro West Orthodontics & Periodontics, La Vista, Nebraska
  - Perio & Implant Associates of Middle TN, Nashville, Tennessee
  - Perio Health Professionals, Houston, Texas
  - Oral Health Specialists, Tacoma, Washington
  - WisNova Institute of Dental Specialists, Kenosha, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jung RE, Pjetursson BE, Glauser R, Zembic A, Zwahlen M, Lang NP. A systematic review of the 5-year survival and complication rates of implant-supported single crowns. Clin Oral Implants Res. 2008 Feb;19(2):119-30. doi: 10.1111/j.1600-0501.2007.01453.x. Epub 2007 Dec 7. PMID 18067597
- [Background] Elani HW, Starr JR, Da Silva JD, Gallucci GO. Trends in Dental Implant Use in the U.S., 1999-2016, and Projections to 2026. J Dent Res. 2018 Dec;97(13):1424-1430. doi: 10.1177/0022034518792567. Epub 2018 Aug 3. PMID 30075090
- [Background] 3. American Dental Association, Patient Smart Dental Implants. Accessed August 15, 2021.
- [Background] Papaspyridakos P, Chen CJ, Singh M, Weber HP, Gallucci GO. Success criteria in implant dentistry: a systematic review. J Dent Res. 2012 Mar;91(3):242-8. doi: 10.1177/0022034511431252. Epub 2011 Dec 8. PMID 22157097
- [Background] Kuhl S, Zurcher S, Mahid T, Muller-Gerbl M, Filippi A, Cattin P. Accuracy of full guided vs. half-guided implant surgery. Clin Oral Implants Res. 2013 Jul;24(7):763-9. doi: 10.1111/j.1600-0501.2012.02484.x. Epub 2012 May 3. PMID 22551385
- [Background] Younes F, Cosyn J, De Bruyckere T, Cleymaet R, Bouckaert E, Eghbali A. A randomized controlled study on the accuracy of free-handed, pilot-drill guided and fully guided implant surgery in partially edentulous patients. J Clin Periodontol. 2018 Jun;45(6):721-732. doi: 10.1111/jcpe.12897. Epub 2018 May 10. PMID 29608793
- [Background] Varga E Jr, Antal M, Major L, Kiscsatari R, Braunitzer G, Piffko J. Guidance means accuracy: A randomized clinical trial on freehand versus guided dental implantation. Clin Oral Implants Res. 2020 May;31(5):417-430. doi: 10.1111/clr.13578. Epub 2020 Jan 31. PMID 31958166
- [Background] 8. ITI.org Consensus Statement, Amsterdam 2018. Implant Placement and Loading Protocols
- [Background] Gallucci GO, Hamilton A, Zhou W, Buser D, Chen S. Implant placement and loading protocols in partially edentulous patients: A systematic review. Clin Oral Implants Res. 2018 Oct;29 Suppl 16:106-134. doi: 10.1111/clr.13276. PMID 30328194
- [Background] Naeini EN, Atashkadeh M, De Bruyn H, D'Haese J. Narrative review regarding the applicability, accuracy, and clinical outcome of flapless implant surgery with or without computer guidance. Clin Implant Dent Relat Res. 2020 Aug;22(4):454-467. doi: 10.1111/cid.12901. Epub 2020 May 13. PMID 32400121
- [Background] Sailer I, Strasding M, Valente NA, Zwahlen M, Liu S, Pjetursson BE. A systematic review of the survival and complication rates of zirconia-ceramic and metal-ceramic multiple-unit fixed dental prostheses. Clin Oral Implants Res. 2018 Oct;29 Suppl 16:184-198. doi: 10.1111/clr.13277. PMID 30328185
- [Background] General Assembly of the World Medical Association. World Medical Association Declaration of Helsinki: ethical principles for medical research involving human subjects. J Am Coll Dent. 2014 Summer;81(3):14-8. PMID 25951678
- [Background] 13. ISO. EN ISO 14155. SS-EN ISO 14155:2011: Swedish Standard Institute; 2011
- [Background] Loe H. The Gingival Index, the Plaque Index and the Retention Index Systems. J Periodontol. 1967 Nov-Dec;38(6):Suppl:610-6. doi: 10.1902/jop.1967.38.6.610. No abstract available. PMID 5237684
- [Background] Geraets W, Zhang L, Liu Y, Wismeijer D. Annual bone loss and success rates of dental implants based on radiographic measurements. Dentomaxillofac Radiol. 2014;43(7):20140007. doi: 10.1259/dmfr.20140007. Epub 2014 Jul 17. PMID 25030551